CLINICAL TRIAL: NCT06413004
Title: Brachyspira and Intestinal Allergy-like Immune Reactions in Patients With Irritable Bowel Syndrome (IBS)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Magnus Simrén (Other)
Responsible Party: Sponsor-Investigator, Magnus Simrén, professor, Sahlgrenska University Hospital
Organization: Sahlgrenska University Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-06370-02
Record Dates: First submitted 2024-05-06; First posted 2024-05-14 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Irritable Bowel Syndrome; Food Sensitivity
Keywords: Irritable Bowel Syndrome; Food Sensitivity; Confocal Laser Endomicroscopy; Colonoscopic Antigen Provocation Test
MeSH Terms: conditions — Irritable Bowel Syndrome; Food Intolerance

STUDY DESIGN:
Intervention Model Description: Unblinded elimination and re-introduction of a positive tested food item, identified during CLE or COLAP
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Positive food item during CLE or COLAP (Other): The food item(s) which were positive during CLE (fluorescein leakage and cell shedding) or COLAP (swelling).
  Interventions: Other: Elimination and re-introduction of CLE or COLAP positive food item(s)

INTERVENTIONS:
Other: Elimination and re-introduction of CLE or COLAP positive food item(s) — Elimination (4 weeks) and re-introduction (4 weeks) of all CLE or COLAP positive food item(s)

SUMMARY:
The aim of this study is to define local immune responses in the GI tract to food antigens in IBS patients, with and without Brachyspira infection, using advanced imaging. We hypothesize that Brachyspira infection can cause IBS symptoms by inducing loss of oral tolerance to dietary antigens through development of food-specific intestinal immune reactions and subsequent development of visceral hypersensitivity.

During this study, the investigators will perform either confocal laser endomiscroscopy (CLE) or colonoscopic antigen provocation test (COLAP) to test to which food items the participants react to. Furthermore, the investigators will perform rectal barostat examination and a sigmoidoscopy without laxatives. The investigators will collect biological samples and the participants will complete several questionnaires.

DETAILED DESCRIPTION:
The aim of this study is to define local immune responses in the GI tract to food antigens in IBS patients with and without Brachyspira infection using advanced imaging. The investigators hypothesize that Brachyspira infection can cause IBS symptoms by inducing loss of oral tolerance to dietary antigens through development of food-specific intestinal immune reactions and subsequent development of visceral hypersensitivity.

Visit 1: inclusion, questionnaires, blood, rectal barostat examination Visit 2: questionnaires, blood, stool, diaries (food and stool), sigmoidoscopy (without laxantives) Allergologist visit (skin prick test and interpretation blood results) Visit 3: stool, confocal laser endomicroscopy (CLE) OR colonoscopic antigen provocation test (COLAP)

Visit 4,5 and 6 only if the CLE or COLAP was positive for (at least) 1 food item

Visit 4: questionnaires and dietician-led instruction which food item to exclude (positive food item(s) during CLE/COLAP), exclusion for 4 weeks Visit 5: questionnaires, stool diary, instructions re-introduction food item(s) Visit 6: questionnaires

QUESTIONNAIRES Baseline questionnaires; demographic, symptoms, symptom/medication/diet history, co-morbid medical conditions

IBS symptoms: IBS-Symptom Severity Scale (IBS-SSS) and Gastrointestinal Symptom Rating Scale (GSRS)-IBS

Psychological distress: Hospital Anxiety and Depression Scale (HADS), Patient Health Questionnaire (PHQ)-9 (both visit 1,4,5,6, generalized Anxiety Disorder 7-item scale (GAD-7)

Somatization: PHQ-15 for the number and severity of bodily symptoms.

Gastrointestinal specific anxiety: Visceral Sensitivity Index (VSI).

Sensitivity: Central Sensitization Inventory (CSI).

Food avoidance and restriction: (ARFID).

Stool habits and GI symptoms: 14-day GI symptom diary based on Bristol Stool Form Scale (BSFS).

Quality of life: IBS-Quality of Life (QOL).

Food intake: 4-days food diary, MealQ.

COLONOSCOPIC ALLERGEN PROVOCATION TEST, COLAP:

* A local allergen provocation test, where dietary antigens (soy, wheat, (egg), gluten and milk), with saline and histamine as negative and positive controls, respectively are injected in the rectosigmoid mucosa (similar to skin prick test used for clinical allergy testing).
* The intestinal reaction is determined visually ("wheal and flare reaction"), and biopsies are taken to characterize the immune response.
* Bowel preparation before the investigation follows the normal clinical routine for colonoscopy, and i.v. sedatives and opioids are given during the investigation according to clinical routines at the endoscopy unit

CONFOCAL LASER ENDOMICROSCOPY, CLE, gastroscopy:

* A probe-based endoscopic technique to study intestinal food reactions after iv injection of fluorescein.
* Disruption of the small intestinal barrier in duodenum upon exposure to food antigens (soy, wheat, egg, gluten, milk, and control) can be determined.

VISCERAL SENSITIVITY:

•Rectal barostat sensitivity measurement: With the rectal barostat, the investigators can measure the rectal sensitivity. A balloon is inserted and inflated in the rectum in a controlled setting. The patient indicates when defined sensory thresholds are reached (first feeling of the balloon, urge to empty bowel, discomfort or pain). When the patient indicates discomfort or pain, or another reason to stop, the balloon inflation will be stopped.

SIGMOIDOSCOPY:

•Flexible sigmoidoscopy without bowel preparation, to interfere as little as possible with the normal gut microenvironment; fresh biopsies for specific analyses and biopsies stored for subsequent analyses.

BIOLOGICAL SAMPLES:

* Blood - and plasma samples: Fasting blood samples are taken for routine blood tests (exclusion of organic diseases) and to determine the metabolic profile and genetic and immunological markers of relevance to intestinal function and nerve function. Serum samples will be analyzed with nuclear magnetic resonance (NMR) for metabolomic profile and microbial composition.
* Fecal - and urine sample: The investigators will characterize the composition and function of the metabolome in detail via 16S analysis, metagenomics, transcriptomics, metabolomics, cell culture and cell count. Urine and fecal samples will also be analyzed with nuclear magnetic resonance (NMR) for metabolomic profile and microbial composition.
* Biopsies (location based on the performed endoscopic examination): The investigators will conduct a detailed analysis of immune cells, proteins, nerve cells, and intestinal bacteria which will allow detailed mapping of intestinal function with respect to nerve, immune and barrier function.

ELIGIBILITY:
Inclusion Criteria:

* Patients with IBS diagnosis according to their treating physician (ROME IV).
* Association between intake of food and GI symptoms.
* Witnessed written informed consent prior to any study procedures.
* Patients who are capable to understand the study and the questionnaires, and to comply with the study requirements.

Exclusion Criteria:

* Patients with relevant concurrent organic GI disease (inflammatory bowel disease, abdominal cancer), or a major disease such as diabetes, uncontrolled thyroid disease, heart disease, kidney disease, liver disease, and active malignant disease (not those that were in remission at least 5 years).
* Patients with a history of bowel surgery (not appendectomy or cholecystectomy) that affects GI motility.
* Patients with systemic food allergy as evidenced by positive allergy tests (blood, prick test).
* Clinical history of severe allergic reactions.
* Patients with concurrent major confounding condition(s) based on the clinician's judgement, e.g. DOMINANT psychiatric disorder, vital depression, alcohol or substance abuse in the last 2 year.
* Female patients who are pregnant or lactating (females of fertile age are requested to use a safe contraceptive) at the time of inclusion.
* Patients who use or used new medications that affect the GI functioning within 1 month before the start of the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-08-03 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
IBS-SSS (Irritable Bowel Syndrom Severity Scoring System) after exclusion (proportion). | 4 weeks after exclusion
  the proportion of participants with an IBS-SSS reduction of ≥50 points, measured before (visit 4) and after (visit 5) exclusion of the CLE or COLAP positive food item(s) (= responders). IBS-SSS: higher IBS-SSS indicate more severe symptoms. Scores ranging 0-500.

SECONDARY OUTCOMES:
IBS-SSS (Irritable Bowel Syndrom Severity Scoring System) after exclusion (absolute) | 4 weeks after exclusion
  IBS-SSS: absolute change of IBS-SSS, measured before (visit 4) and after (visit 5) EXCLUSION of the CLE or COLAP positive food item(s). Higher IBS-SSS indicate more severe symptoms. Scores ranging 0-500.
IBS-SSS (Irritable Bowel Syndrom Severity Scoring System) after reintroduction (proportion) | 4 weeks after reintroduction
  IBS-SSS: the proportion of participants with an IBS-SSS increase of ≥50 points, measured before (visit 5) and after (visit 6) the REINTRODUCTION of the CLE or COLAP positive food item(s): responders vs non-responders (as based on the primary outcome). Higher IBS-SSS indicate more severe symptoms. Scores ranging 0-500.
IBS-SSS (Irritable Bowel Syndrom Severity Scoring System) after reintroduction (absolute) | 4 weeks after reintroduction
  IBS-SSS: the absolute change of IBS-SSS, measured before (visit 5) and after (visit 6) the REINTRODUCTION of the CLE or COLAP positive food item(s): total group and responders vs non-responders (as based on the primary outcome)
GSRS-IBS (the Gastrointestinal Symptom Rating Scale Irritable Bowel Syndrome version) after exclusion | 4 weeks after exclusion
  change of total and subscores before (visit 4) and after (visit 5) EXCLUSION of the CLE or COLAP positive food item(s). Total group and responders vs non-responders (as based on the primary outcome). Higher GSRS-IBS indicate more severe symptoms. After calculating of the average scores, those range 1-7.
GSRS-IBS (the Gastrointestinal Symptom Rating Scale Irritable Bowel Syndrome version) after reintroduction | 4 weeks after reintroduction
  change of total and subscores before (visit 5) and after (visit 6) REINTRODUCTION of the CLE or COLAP positive food item(s). Total group and responders vs non-responders (as based on the primary outcome). Higher GSRS-IBS indicate more severe symptoms. After calculating of the average scores, those range 1-7.
HAD (Hospital Anxiety and Depression scale) after exclusion | 4 weeks after exclusion
  change of total and subscores before (visit 4) and after (visit 5) EXCLUSION of the CLE or COLAP positive food item(s). Total group and responders vs non-responders (as based on the primary outcome). Higher HAD scores indicate more symtoms of anxiety and depression. Total score ranging 0-42 and the two subscores (anxiety and depression) ranging 0-21.
HAD (Hospital Anxiety and Depression scale) after reintroduction | 4 weeks after reintroduction
  change of total and subscores before (visit 5) and after (visit 6) REINTRODUCTION of the CLE or COLAP positive food item(s). Total group and responders vs non-responders (as based on the primary outcome). Higher HAD scores indicate more symtoms of anxiety and depression. Total score ranging 0-42 and the two subscores (anxiety and depression) ranging 0-21.
PHQ12 (the Patient Health Questionnaire - 12) after exclusion | 4 weeks after exclusion
  change of scores before (visit 4) and after (visit 5) EXCLUSION of the CLE or COLAP positive food item(s). Total group and responders vs non-responders (as based on the primary outcome). Higher PHQ12 scores indicate more bothersome non-GI somatic symptoms. Scores ranging 0-24, with a subanalysis excluding mentrual problems, leading to a range 0-22.
PHQ12 (the Patient Health Questionnaire - 12) after reintroduction | 4 weeks after reintroduction
  change of scores before (visit 5) and after (visit 6) REINTRODUCTION of the CLE or COLAP positive food item(s). Total group and responders vs non-responders (as based on the primary outcome). Higher PHQ12 scores indicate more bothersome non-GI somatic symptoms. Scores ranging 0-24, with a subanalysis excluding mentrual problems, leading to a range 0-22.

CONTACTS AND LOCATIONS:
Locations (1):
- Mag-tarmlab, Dept of Internal Medicine, Sahlgrenska University Hospital, Gothenburg, Sweden

DOCUMENTS (1):
  • Study Protocol (2024-04-29): https://cdn.clinicaltrials.gov/large-docs/04/NCT06413004/Prot_000.pdf